CLINICAL TRIAL: NCT05410275
Title: Chronic Anticoagulation in End-stage Renal Disease Patients: Pharmacokinetics and Pharmacodynamic of a Reduced Dose Regimen of Rivaroxaban
Brief Title: Chronic Anticoagulation With a Reduced Dose Regimen of Rivaroxaban in End-stage Renal Disease Patients
Acronym: CARD-AXA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR190242-CARD-AXA
Record Dates: First submitted 2022-02-02; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hemodialysis Patients
Keywords: Kidney Diseases; Therapeutic drug monitoring
MeSH Terms: conditions — Kidney Diseases | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rivaroxaban (Experimental): Rivaroxaban 5 mg daily, administered orally, during 3 consecutive days. After a wash-out period of 4 days, Rivaroxaban 10 mg daily, administered orally, during 3 consecutive days.
  After a wash-out period of 4 days, Rivaroxaban 15 mg daily, administered orally, during 3 consecutive days.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Experimental group Each patient will receive successively over 3 distinct periods the 3 doses of rivaroxaban to be evaluated, i.e., 5 mg, 10 mg, and 15 mg as a single daily dose (once daily over 3 days for each dose).

SUMMARY:
Atrial fibrillation is the most frequent cardiac rhythm disorder and its prognosis is essentially marked by the risk of embolic events. Its treatment is based on long-term oral anticoagulant therapy according to the risk of embolic events assessed by risk scores such as the CHA2DS2-Vasc score, but this prescription is associated with a risk of hemorrhagic events that must be taken into consideration when deciding on the treatment for a given patient. There are two categories of validated oral anticoagulant treatments for the prevention of embolic events in atrial fibrillation: antivitamin K agents, which have long been the reference treatment but are restrictive and difficult to use because of a narrow therapeutic window, and direct oral anticoagulants, which are now the first-line treatment but have not been evaluated in phase II and III studies in patients with severe renal failure. End-stage renal disease (clearance <15 mL/min/1.73m2), particularly at the dialysis stage, is a risk factor for cardiovascular disease in its own right, and a significant number of patients develop atrial fibrillation. Given the co-morbidities associated with renal failure, in particular hypertension, patients with renal failure undergoing dialysis and suffering from atrial fibrillation are generally at a higher risk of embolism than patients without renal failure, but also at a higher risk of bleeding. Thus, if the indication for prescribing oral anticoagulant therapy is clear in this population, the associated bleeding complications are also more frequent and more serious in these patients who have regular vascular accesses in the context of hemodialysis. There is thus a real need for reliable therapeutic alternatives with a better benefit/risk ratio than antivitamins K.

Translated with www.DeepL.com/Translator (free version)

DETAILED DESCRIPTION:
Chronic dialysis patients are a special population because the constraints linked to their disease (3 dialyses per week) make them a captive population that nephrologists know perfectly well. If the identification of the subjects to be included does not pose any problem, it is more their adherence to the project which is likely to be more difficult because it implies additional constraints in these patients with potentially many comorbidities.

This proof-of-concept study will identify the dose of rivaroxaban with the best pharmacokinetic/ pharmacodynamic profile in chronic hemodialysis patients. It will then be possible to envisage a larger study of the type of a national Hospital Clinical Research Program (PHRC) in order to evaluate the dose of rivaroxaban chosen in hemodialysis patients with atrial fibrillation with an indication for oral anticoagulation on the basis of morbidity-mortality criteria in comparison with treatment with antivitamins K that is well conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years of age,
* Chronic hemodialysis patient for at least 3 months,
* Affiliated or beneficiary of a social security plan,
* Having signed a written and informed consent.

Exclusion Criteria:

* Any indication for long-term oral anticoagulation (atrial fibrillation, venous thromboembolic disease, mechanical valve prostheses, intracardiac thrombosis, etc.)
* Double anti-platelet aggregation for any reason or an aspirin dose greater than 160 mg/day
* Uncontrolled hypertension (BP > 180/110 mmHg)
* Ischemic stroke within 30 days prior to inclusion
* History of major unprovoked hemorrhage (leading to hospitalization or transfusion) regardless of age
* Surgery within 30 days prior to inclusion
* High-risk bleeding condition in addition to renal failure (such as known coagulation disorder, thrombocytopenia (< 100G/L), active neoplasia of the digestive or urinary tract, or presence of intracranial vascular malformation)
* Severe hepatic impairment
* Use of strong CYP3A4 inducers, including rifampin, St. John's Wort, carbamazepine, phenytoin, phenobarbital
* Non-compliant patients
* Pregnant or breastfeeding women, women of childbearing age without effective contraception
* Contraindication to the administration of an anticoagulant treatment such as anti-phospholipid antibody syndrome
* Known allergy to rivaroxaban or to one of its excipients (lactose monohydrate)
* Patients under guardianship or conservatorship
* Patients already participating in an ongoing study or who have participated in a study that ended less than 30 days prior to the inclusion date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics of 3 reduced dose regimen of rivaroxaban (5 mg/day, 10 mg/day, or 15 mg/day) | 1 month
  Plasma anti-Xa activity assessment (international unit per milliliter, IU/mL) on serial blood sampling at specified time points
Pharmacokinetics of 3 reduced dose regimen of rivaroxaban (5 mg/day, 10 mg/day, or 15 mg/day) | 1 month
  Direct measurement of Rivaroxaban plasma level (nanogram per milliliter, ng/mL) on serial blood sampling at specified time points

SECONDARY OUTCOMES:
Hemorrhagic risk assessment of 3 reduced dose regimen of rivaroxaban (5 mg/day, 10 mg/day, or 15 mg/day) | 1 month
  Every bleeding event will be reported and classified according to the BARC classification

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice IVANES, MD-PhD, Study Director — University Hospital of TOURS